CLINICAL TRIAL: NCT06065696
Title: Compliance With Enhanced Recovery After Surgery Protocol on Early Mobilization After Colorectal Surgery in Tertiary Hospital in Indonesia
Brief Title: Enhanced Recovery After Surgery Protocol on Early Mobilization After Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aldy Heriwardito, Principal Investigator, Indonesia University
Other Study IDs: IndonesiaUAnes112
Record Dates: First submitted 2023-07-31; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Enhanced Recovery After Surgery; Anesthesia; Surgery-Complications; Colorectal; Early Mobilization
Keywords: early mobilization; Enhanced Recovery After Surgery; PONV prophylaxis; fluid management; pain management
MeSH Terms: conditions — Agnosia | interventions — Early Ambulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early mobilization: Patients who achieved early mobilization after colorectal surgery
  Interventions: Procedure: Early mobilization
- No early mobilization: Patients who did not achieve early mobilization after colorectal surgery
  Interventions: Procedure: No early mobilization

INTERVENTIONS:
Procedure: Early mobilization — Patients who received early mobilization in postoperative period
  Groups: Early mobilization
Procedure: No early mobilization — Patients who did not receive early mobilization in postoperative period
  Groups: No early mobilization

SUMMARY:
Early mobilization is an important factor in increasing postoperative colorectal surgeries outcome. There are four components held by anesthesiologist in Enhanced Recovery After Surgery protocol for colorectal surgery in our hospital: post operative nausea and vomiting (PONV) prophylaxis, intraoperative fluid management, intraoperative multimodal analgesia, and postoperative opioid-free pain management. Although early mobilization affected by postoperative pain, vomiting and nausea, and fluid balance management, nonetheless, there is no clear evidence of how much each of these components will affect early mobilization.

DETAILED DESCRIPTION:
Early mobilization is an important factor in increasing postoperative colorectal surgeries outcome. There are four components held by anesthesiologist in ERAS protocol for colorectal surgery in our hospital: PONV prophylaxis, intraoperative fluid management, intraoperative multimodal analgesia, and postoperative opioid-free pain management. Although early mobilization affected by postoperative pain, vomiting and nausea, and fluid balance management, nonetheless, there is no clear evidence of how much each of these components will affect early mobilization. This study was a retrospective cohort study by collecting secondary data from patients underwent elective colorectal surgery in our hospital from January 2020 to December 2022. The outcomes assessed were early mobilization rate and factors affecting it (PONV prophylaxis, intraoperative fluid management, intraoperative multimodal analgesia, and postoperative opioid-free pain management).

ELIGIBILITY:
Inclusion criteria

* Patient underwent colorectal surgery in Cipto Mangunkusumo Hospital from 2020 to 2022
* Age 18-60 years old
* American Society of Anesthesiologist (ASA) physical status 1, 2, and 3

Exclusion criteria

* Patients who were not intubated on postoperative period
* Patients who had physical limitation during preoperative mobility test

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients underwent colorectal surgery in Cipto Mangunkusumo Hospital during 2020 to 2022
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Early mobilization | Within 24 hours after surgery
  Number of patients who can walk within 24 hours after surgery
PONV prophylaxis | Given during intraoperative period
  Number of patients who received prophylaxis given for PONV
Multimodal analgesia | Given during intraoperative period
  Number of patients who got multimodal analgesia, which consists of epidural anesthesia or peripheral nerve block
Intraoperative fluid management | Given during intraoperative period
  Number of patients who achieved fluid balance of zero or near zero
Postoperative pain management | Immediately after surgery until discharge, assessed until hospital discharge, up to 50 days
  Number of patients who received postoperative pain management without opioid

CONTACTS AND LOCATIONS:
Overall Officials: Aldy Heriwardito, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No